CLINICAL TRIAL: NCT03245645
Title: FODMAP Reintroduction in Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Lin Chang, MD, Director, Digestive Health and Nutrition Clinic, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16-000934
Record Dates: First submitted 2017-07-25; First posted 2017-08-10 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Irritable Bowel Syndrome With Diarrhea; Irritable Bowel Syndrome With Mixed Bowel Habits
Keywords: FODMAP; IBS; Diet; Re-introduction; Fructose
MeSH Terms: interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 100% Fructose (Experimental): The fructose group will help to determine whether an absolute amount of fructose will lead to IBS symptoms.
  Interventions: Other: Dietary Intervention
- 100% Glucose (Placebo Comparator): The glucose group will serve as a control since glucose is not a FODMAP and as a result is not expected to lead to recurrent symptoms.
  Interventions: Other: Dietary Intervention
- Fructose and Glucose (Active Comparator): The glucose/fructose mixture group is a cross comparison group that will determine whether the relative excess fructose concentration is an important cause of IBS symptoms.
  Interventions: Other: Dietary Intervention

INTERVENTIONS:
Other: Dietary Intervention — Food may be linked to changes in motility, visceral sensation, gut microbiome, intestinal permeability, immune activation and brain-gut axis. This study will focus on fructose, which is one of the main components of FODMAP (Fermentable oligosaccharides, dissacharides, mono-saccharides and polyols) foods. Fructose is a common part of the Western diet and can be consumed as a free monosaccharide, part of sucrose, or in polymers referred to as fructans. FODMAP foods are thought to induce gastrointestinal symptoms including gas, bloating, abdominal pain or discomfort, and loose stools by increasing small bowel water content and increasing gas production by fermentation of foods by gut bacteria. Studies including a recent controlled clinical trial demonstrated that a low FODMAP diet can be an effective nutritional therapy.

SUMMARY:
The purpose of this study is to determine the amount and timing of when certain Fermentable Oligo-Di-Monosaccharides and Polyols (FODMAPs), specifically fructose, can be safely reintroduced into the diet of Irritable Bowel Syndrome (IBS) patients that have successfully completed a low-FODMAP elimination diet. The FODMAP diet is an effective treatment for IBS; however it is unclear how patients can successfully reintroduce and liberalize fructose into their diet. The low FODMAP diet is thought to reduce IBS symptoms by decreasing water content and gas production in the bowel and also possibly by altering gut bacteria. Although use of the FODMAP elimination diet can initially successfully treat IBS symptoms for up to 50-75% of patients, the reintroduction diet is difficult for patients to complete and maintain for long periods of time because current methods for reintroduction of FODMAPs are imprecise leading to frequent recurrent symptoms. As a result, patients often continue the low FODMAP elimination diet for additional months because they have difficulties knowing how to add back FODMAPs into their diet. There are no studies to date to help guide patients with FODMAP reintroduction.

DETAILED DESCRIPTION:
Research supports clinical experience that ingestion of food often triggers the emergence or exacerbation of symptoms in the majority of patients with irritable bowel syndrome (IBS). While IBS remains primarily a symptom driven entity, our understanding of its pathophysiology is evolving. However, comparatively little research has focused on the specific role of certain foods and how they prompt the development of IBS symptoms.

Food may be linked to changes in motility, visceral sensation, gut microbiome, intestinal permeability, immune activation and brain-gut axis. This study will focus on fructose, which is one of the main components of FODMAP (fermentable oligosaccharides, disacharides, mono-saccharides and polyols) foods. Fructose is a common part of the Western diet and can be consumed as a free monosaccharide, part of sucrose, or in polymers referred to as fructans. There are no human gut specific fructose transporters. Rather glucose transporters are used (GLUT 2,5) leading some to hypothesize that over ingestion of these agents may trigger some of the enteric complaints of patients with IBS. The literature on fructose malabsorption gives varying threshold amounts: from 15 to 50 grams in healthy controls, and from 5 to 50 grams in IBS patients/known malabsorbers (Barrett, 2007; Rao, 2007; Frieling, 2011). Average daily fructose consumption in the American diet is approximately 34 grams, with a range of 15 to 54 grams, which falls well within the threshold levels (Frieling, 2011). FODMAP foods are thought to induce gastrointestinal symptoms including gas, bloating, abdominal pain or discomfort, and loose stools by increasing small bowel water content and increasing gas production by fermentation of foods by gut bacteria. Studies including a recent controlled clinical trial demonstrated that a low FODMAP diet can be an effective nutritional therapy.

There are risks to prolonged use of a low FODMAPs diet. A study from 2012 suggested that continued restriction of FODMAPS (longer than 4 weeks) can lead to reduction of luminal bifidobacteria in patients with IBS. Bifidobacteria mainly inhabit the large intestine where they produce short chain fatty acids (SCFA) as byproducts, including butyrate, shown to be important for colorectal cancer prevention and limit enteropathogenic colonization. Furthermore the diet is very restrictive and difficult for patients to maintain over time.

However, important clinical questions include when FODMAPS can be safely reintroduced into the diet, how quickly this can be accomplished, and what is a daily threshold of intake that is acceptable for IBS patients who respond or do not respond to a low FODMAPs diet. There are no evidence based answers to these questions, and it is in this setting that we propose our current project.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18+ years or older) with a diagnosis of IBS-D or IBS-M based on Rome IV criteria
* Diarrhea must occur 2 or more days per week
* Patients on current pharmacological therapy for their gastrointestinal complaints can enroll in the study as long as they have been on a stable dose for at least 30 days.

Exclusion Criteria:

* Significant comorbidities that are associated with GI symptoms (e.g. diabetes, scleroderma, SLE), history of GI surgery excluding appendectomy, or prior organic GI illness
* Antibiotics taken in the past 2 months
* Current disordered eating patterns (diagnosed eating disorder; as per verbal ESP questionnaire)
* Current history of greater than moderate alcohol intake (more than 1 drink per day for women, more than 2 drinks per day for men, binge drinking behavior of 5+ drinks in a single session once per week)
* Cannot have had a cholecystectomy in the past 6 months prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-03-24 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Adequate relief of IBS symptoms in past 7 days | Baseline, 4 weeks (post-elimination diet)
  As indicated by the study coordinator asking the participant "Have you had adequate relief of your IBS symptoms in the past 7 days?"
Highest amount of grams of sugar in solutions that do not significantly increase IBS symptoms | Daily, during weeks 5-7 (reintroduction phase)
  As measured by 100 MM Visual Analog Scale (VAS) with 0 representing no symptoms for overall gastrointestinal symptoms.

SECONDARY OUTCOMES:
Change in IBS-symptom severity scale | Baseline, 4 weeks (post-elimination diet), 7 weeks (post-reintroduction phase)
  This is a validated symptom questionnaire pertaining to irritable bowel syndrome symptoms
Change in Visceral Sensitivity Index (VSI) | Baseline, 4 weeks (post-elimination diet), 7 weeks (post-reintroduction phase)
  This is a self-report measure of the gastrointestinal symptom-specific anxiety (GSA) of patients with irritable bowel syndrome (IBS)
Change in Personal Health Questionnaire (PHQ-15) | Baseline, 4 weeks (post-elimination diet), 7 weeks (post-reintroduction phase)
  This is a validated symptom questionnaire pertaining to somatic symptoms severity
Change in abdominal pain severity | Baseline, 4 weeks (post-elimination diet), 7 weeks (post-reintroduction phase)
  This is a self-report measure of the severity of abdominal pain during the week before report gathered by circling a number from 0-20 with 20 being the most intense pain imaginable.
Change in overall severity of gastrointestinal symptoms | Baseline, 4 weeks (post-elimination diet), 7 weeks (post-reintroduction phase)
  This is a self-report measure of the overall severity of gastrointestinal symptoms during the week before report gathered by circling a number from 0-20 with 20 being the most intense symptoms imaginable.
Change in severity of the sensation of bloating, abdominal fullness or visible distension | Baseline, 4 weeks (post-elimination diet), 7 weeks (post-reintroduction phase)
  This is a self-report measure of the severity of the sensation of bloating, abdominal fullness, or visible distension in the patient's belly that the patient has experienced during the week before report gathered by circling a number from 0-20 with 20 being the most intense sensation imaginable.
Change in intestinal microbiota | Baseline, 4 weeks (post-elimination diet)
  This is a measure of the intestinal microbiota 16S rRNA gene signatures in the patients' stool before and after the low FODMAP diet.
Change in visceral sensitivity index score | Baseline, 4 weeks (post-elimination diet), 7 weeks (post-reintroduction phase)
  This is a validated symptom questionnaire pertaining to gastrointestinal symptom related anxiety in patients with irritable bowel syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Chang, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States